CLINICAL TRIAL: NCT02767466
Title: A Preliminary Study on Acute Affective Responses Focussing on Differences Between Physical Therapy and Robotic Assisted Gait Training
Brief Title: Affective Responses in Neurological Rehabilitation
Status: Completed | Type: Observational
Sponsor: Universitaet Innsbruck (Other)
Responsible Party: Principal Investigator, Martin Burtscher, Prof Martin Burtscher, Universitaet Innsbruck
Other Study IDs: APTRAGT001
Record Dates: First submitted 2016-04-22; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Neurological Incidents; Stroke; Traumatic Brain Injury
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- G: All participants were randomly exposed to two different treatments:
  * Conventional physical therapy (no specific device used)
  * Robotic assisted gait training (Lokomat, Hocoma AG, Switzerland)
  We consider the study as observational, since the both interventions of the study (physical therapy, robotic assisted gait training) did not change in the patients' usual therapy plan, as they received both interventions daily.
  We only added diagnostic interventions to assess the affective responses.
  Interventions: Procedure: Physical therapy and robotic assisted gait training

INTERVENTIONS:
Procedure: Physical therapy and robotic assisted gait training

SUMMARY:
Using a single blind within-subject design, 16 patients with neurological disorders were randomly exposed to two different treatments: physical therapy and robotic assisted gait training. Both before and after the treatments, a self-report Mood Survey Scale (MSS) was used to assess the effects on the treatment on distinct affective states. The subscales of the MSS were tested for pre-post changes and different effects between treatments with non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation
* neurological incident

Exclusion Criteria:

* lack of communication ability
* interference of consciousness
* inability to speak German language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological disorders
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change of subscales of mood survey scale from pre to post treatment | 30-60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kopp, Prof, Study Director — Univeryity of Innsbruck